CLINICAL TRIAL: NCT02815917
Title: Evaluation of D3 Receptor Occupancy Using [18F]FLUORTRIOPRIDE ([18F]FTP) PET/CT
Brief Title: Evaluation of D3 Receptor Occupancy Using FLUORTRIOPRIDE ([18F]FTP) PET/CT
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 824853
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: D3 Dopamine Receptor; Cocaine-dependent; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1a: Lorazepam; 1b: Perphenazine (Experimental): Up to 5 healthy volunteers will participate in a double-blind, placebo controlled serial imaging cohort 1a. Each subject will undergo two dynamic [18F]FTP PET/CT brain scans on two separate days. On one scan day the patient will receive an IV injection of normal saline (placebo) prior to the FTP brain scan, on the other scan day the patient will receive an IV injection of lorazepam prior to the planned FTP injection scan. The type of injection (placebo versus lorazepam) will be double-blinded to the patient and the injecting nuclear medicine Authorized User. Up to 5 subjects will participate in Cohort 1b where subjects will undergo two FTP PET/CT with and without perphenazine.
  Subjects in all cohorts are required to have a structural brain MRI performed within 1 year of study enrollment. If the subject has not had a brain MRI that is deemed acceptable for use for this study, they will be asked to undergo a research brain MRI after they have consented for this study.
  Interventions: Drug: [18F]FTP PET/CT
- Cohort 2: Healthy Volunteer Test/Retest (Experimental): Up to 10 healthy volunteers will participate in a serial imaging cohort. Each subject will undergo two dynamic [18F]FTP PET/CT brain scans on two separate days.
  Subjects in all cohorts are required to have a structural brain MRI performed within 1 year of study enrollment. If the subject has not had a brain MRI that is deemed acceptable for use for this study, they will be asked to undergo a research brain MRI after they have consented for this study.
  Interventions: Drug: [18F]FTP PET/CT
- Cohort 3: Arterial sampling (Experimental): Up to 5 cocaine-dependent males who are voluntarily seeking treatment for cocaine dependence will participate in this imaging cohort. Each subject will undergo one dynamic [18F]FTP PET/CT brain scan. Patients will have an arterial line placed for blood draws during the scan. This group will be used to determine the arterial blood input and FTP parent to metabolite ratio curves for FTP for a cocaine-dependent patient population for comparison with previously collected data in healthy normal volunteers.
  Subjects in all cohorts are required to have a structural brain MRI performed within 1 year of study enrollment. If the subject has not had a brain MRI that is deemed acceptable for use for this study, they will be asked to undergo a research brain MRI after they have consented for this study.
  Interventions: Drug: [18F]FTP PET/CT
- Cohort 4: Cocaine-dependent Test/Retest (Experimental): Up to 5 cocaine-dependent males who are voluntarily seeking treatment for cocaine dependence will participate in this imaging cohort. Each subject will undergo two dynamic [18F]FTP PET/CT brain scans on two separate days. This group will be used to test the variability of the [18F]FTP uptake measures in cocaine-dependent patients when scans are done following the consistent procedures with no other interventions.
  Subjects in all cohorts are required to have a structural brain MRI performed within 1 year of study enrollment. If the subject has not had a brain MRI that is deemed acceptable for use for this study, they will be asked to undergo a research brain MRI after they have consented for this study.
  Interventions: Drug: [18F]FTP PET/CT

INTERVENTIONS:
Drug: [18F]FTP PET/CT — All PET/CT imaging sessions will include an injection of [18F]FTP. Pilot data will be collected to evaluate preliminary information on brain uptake of [18F]FTP in healthy volunteers and cocaine-dependent volunteers.

SUMMARY:
Preclinical work suggests that D3 dopamine receptors may be important in the study of the pathophysiology of affective disorders, psychotic disorders and addiction. D3 receptors may also play a role in dystonia, Parkinson's disease and response to treatment of these disorders. However, there has been a lack of specific radioligands for imaging D3 receptors. This proposed protocol will evaluate the uptake of [18F]FTP as a more specific in vivo measure of D3 receptor binding in the brain in healthy volunteers subjects after injection of lorazepam vs placebo, and in cocaine-dependent subjects. Test-retest scans will evaluate the variability of [18F]FTP uptake measures in both healthy volunteer subjects and cocaine-dependent subjects.

ELIGIBILITY:
Inclusion Criteria for Cohort 1 and 2 (Healthy Volunteers):

1. Participants will be 18-60 years of age
2. "Healthy volunteer" is defined as being in good general health in the opinion of an investigator (controlled diabetes, controlled hypertension or other well controlled chronic medical conditions may be allowed at the discretion of an investigator if they do not believe they will increase patient risk or interfere with the collection of imaging data; specific excluded conditions are described under exclusion criteria)
3. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria for Cohort 1 and 2 (Healthy Volunteers)

1. Females who are pregnant at the time of screening will not be eligible for this study, urine pregnancy test will be performed in women of child-bearing potential at screening.
2. History of contraindications to lorazepam (sensitivity to diazepines, sleep apnea syndrome or severe respiratory insufficiency) as assessed by medical record review and/or self-reported
3. History of significant gallbladder, kidney or liver disease as assessed by medical record review and/or self-reported OR total bilirubin > 1.5 x ULN, ALT or AST > 3 x ULN or creatinine clearance estimated to be less than 60 ml/min at screening. Subjects with history of cholecystectomy will not be excluded.
4. History of epilepsy or seizure disorder as assessed by medical record review and/or self-reported
5. History of head trauma, that in the opinion of an investigator may interfere with the uptake of [18F]FTP as assessed by medical record review and/or self-reported
6. History of Post-Traumatic Stress Disorder (PTSD), bipolar disorder, schizophrenia or psychotic disorder, or substance use disorders, as assessed by medical record review and/or self-reported
7. Use of dopaminergic CNS stimulants (prescription, over-the counter or recreational drugs) within 30 days of screening intake visit, as assessed by review of health history form and concomitant medication review at screening intake visit (from medical record and/or self-reported) that are deemed by a physician investigator to have a potential influence on the binding of [18F]FTP
8. Positive urine drug screen at the screening intake visit
9. Self-reported current alcohol consumption that exceeds greater than 25 drinks per week
10. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
11. Participants with self-reported current nicotine dependence will be excluded. Participants with self-reported history of nicotine use but who report no use within at least 3 months prior to study enrollment will be eligible for the study if they have a negative urine dipcard test for nicotine/cotinine at screening.

Inclusion criteria for Cohort 3 and 4 (cocaine-dependent)

1, Participants will be males 18-60 years of age 2. Cocaine-dependent (moderate to severe cocaine use disorder, based on DSM-5 criteria), voluntarily seeking treatment for cocaine dependence 3. Smoking is they self-reported primary route of cocaine administration 4. In the past 30 days, no less than $100-worth of cocaine was used by self-report 5. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion criteria for Cohort 3 and 4 (cocaine-dependent)

1. Meets DSM-5 criteria for moderate to severe substance use disorder for any substance other than cocaine, alcohol, marijuana or nicotine as determined by semi-structured interview. Patients with comorbid alcohol use disorder will be accepted if their alcohol use disorder is not severe enough to require a medicated alcohol detoxification per standard UPHS policies
2. History of significant gallbladder, kidney or liver disease as assessed by medical record review and/or self-reported OR total bilirubin > 1.5 x ULN, ALT or AST > 3 x ULN or creatinine clearance estimated to be less than 60 ml/min at screening. Subjects with history of cholecystectomy will not be excluded.
3. History of epilepsy or seizure disorder as assessed by medical record review and/or self-reported
4. History of head trauma, that in the opinion of an investigator may interfere with the uptake of [18F]FTP as assessed by medical record review and/or self-reported
5. History of Post-Traumatic Stress Disorder (PTSD), bipolar disorder, schizophrenia or psychotic disorder as assessed by medical record review and/or self-reported. History of unipolar depression or anxiety disorder may be accepted; current depression or anxiety may be accepted if the severity does not require psychoactive medication.
6. Currently requires treatment with any psychoactive medications
7. Any current medical condition, psychiatric disorder, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assess the difference in uptake [18F]fluortriopride in D3-rich regions in the brain after injection of lorazepam versus placebo in healthy volunteers | 2 years
Measure test-retest variability of [18F]fluortriopride uptake measures in healthy volunteer subjects and cocaine-dependent subjects | 2 years
Evaluate uptake of [18F]fluortriopride in D3-rich areas of the brain in cocaine-dependent volunteers and compare to uptake in healthy volunteer subjects | 2 years

SECONDARY OUTCOMES:
Correlate standard measures of cocaine craving and withdrawal to [18F]FTP uptake in cocaine-dependent subjects | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Dubroff, MD PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No